CLINICAL TRIAL: NCT00000269
Title: Pergolide Treatment for Substance Abusers
Brief Title: Pergolide Treatment for Substance Abusers - 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York State Psychiatric Institute (Other)
Purpose: Treatment
Other Study IDs: NIDA-09236-4; P50-09236-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Pergolide

INTERVENTIONS:
Drug: Pergolide

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pergolide for cocaine dependence.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1995-10; Study Completion 2001-12

PRIMARY OUTCOMES:
Side effects
Craving
Drug use
Improvement in functioning
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kleber, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States